CLINICAL TRIAL: NCT03869008
Title: Potential Benefit for Non Invasive Vagus Nerve Stimulation (nVNS) Using GammaCore in the Treatment of Raynaud's Phenomena.
Brief Title: Potential Benefit for Non Invasive Vagus Nerve Stimulation Using GammaCore in the Treatment of Raynaud's Phenomena.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding is no longer available
Sponsor: University of Toledo Health Science Campus (Other)
Collaborators: ElectroCore INC (Industry)
Responsible Party: Principal Investigator, Bashar Kahaleh, M.D, Professor of Medicine, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: gammaCore RP
Record Dates: First submitted 2019-02-20; First posted 2019-03-11 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-05

CONDITIONS: Raynaud Phenomenon; Primary Raynaud Phenomenon; Raynaud Disease; Raynaud Syndrome
MeSH Terms: conditions — Raynaud Disease

STUDY DESIGN:
Intervention Model Description: At randomization subjects are randomized to 2 groups, the Experimental group and the Sham group.
  The Experimental group will use the study device from randomization to the end of the study.
  The Sham group will use the Sham device for 4 weeks after randomization then be switched to the study device for the rest of the study.
Who Masked: Participant
Masking Description: Subjects randomized to the Experimental group will use the gammaCore Sapphire till the end of the study. Subjects in this group will become un-blinded in the open label phase of the study at 4 weeks after randomization.
  Subjects randomized to the Sham group will use the Sham device for 4 weeks. Subjects in the Sham group will become un-blinded in the open label phase of the study at 4 weeks after randomization and be switch to the gammaCore Sapphire for the rest of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham Device Group (Sham Comparator): 15 patients will be randomized to the Sham device for the first half of the treatment window then switch to the gammaCore Sapphire device (study device) for the rest of the study.
  The Sham device will look exactly like the gammaCore Sapphire device but will not deliver non invasive vagus nerve stimulation.
  Interventions: Device: gammaCore Sapphire; Device: Sham Device
- gammaCore Sapphire (Study Device) Group (Experimental): 15 patients will be randomized to the gammaCore Sapphire device for the full length of the treatment window.
  Interventions: Device: gammaCore Sapphire

INTERVENTIONS:
Device: gammaCore Sapphire — gammaCore SapphireTM (non-invasive vagus nerve stimulator) is intended to provide non-invasive vagus nerve stimulation (nVNS) on the side of the neck. gammaCore provides a mild electrical stimulation to the vagus nerve, which runs through the neck and carries information to the central nervous system.
  Subjects will be instructed to use the gammaCore Sapphire to stimulate 2 minutes on each side of the neck, twice a day, every day. The subject controls the intensity level of the electrical stimulation.
Device: Sham Device — The Sham device delivers no electrical stimulations but subjects randomized to the Sham device will received the same instructions to use the Sham device to stimulate 2 minutes on each side of the neck, twice a day, every day for the first 4 weeks after randomization.
  Arms: Sham Device Group

SUMMARY:
Raynaud's phenomenon (RP) is a common vascular disorder that affects approximately 10% of the general population. RP is associated with significant morbidity that may include loss of the digits due to repeated episodes of vasospasm of the digital arteries in addition to significant impairment of quality of life. It is well known that cold exposure precipitates episodes of RP, but the mechanism for cold sensitivity is not known, and treatment of RP is not satisfactory to the patients and their physicians.

The goal in this study is to test the possibility that non invasive vagus nerve stimulation (nVNS) with gammaCore which is already approved by the FDA for headaches and migraines may be an effective and well tolerated therapy for Raynaud's Phenomenon.

DETAILED DESCRIPTION:
Raynaud's phenomenon (RP) is a common vascular disorder that that affects approximately 10% of the general population. RP causes some areas of the body (i.e. fingers and toes) to feel cold and numb in response to cold exposure or emotional stress. Raynaud's phenomenon is characterized by reversible vasospasm of the fingers and toes. This reversible narrowing of the small arteries induces episodes of color changes of the fingers and toes. During an attack of Raynaud's, affected areas of the skin usually first turn white, then they often turn blue and feel cold and numb (pins and needles). As the fingers warm and circulation improves the affected areas may turn red, throb and tingle.

Moreover, Raynaud's phenomenon can be associated with significant morbidity that may include ulceration of fingers and loss of the fingers and toes due to repeated episodes of reversible narrowing of arteries supplying blood to the finger and toes. It is well known that cold exposure leads to episodes of RP, but the mechanism for cold sensitivity is not known, and treatment of RP is not satisfactory to the patients and their physicians.

Raynaud's phenomenon is classified as Primary Raynaud's phenomenon (PRP) in the absence of other vascular or connective tissue disease. Raynaud's phenomenon is classified as Secondary Raynaud's phenomenon (SRP) if it is associated with connective tissue disease, like systemic sclerosis (SSc, Scleroderma).

Treatment of Raynaud's phenomenon is not satisfactory in general, as current therapy employing calcium channel blockers and other vasodilators are frequently ineffective or not well tolerated, due to significant side effects.

Noninvasive vagus nerve stimulation (nVNS) is currently FDA approved for therapeutic uses in patient ages 12 and above to treat cluster and migraine headaches. Recent studies have shown that vagal nerve stimulation has vasodilatory and anti-inflammatory properties which has led to more preclinical research examining vagus nerve stimulation as treatment for a wider range of inflammatory and autoimmune disorders. Vagus nerve stimulation has shown promising results in treating chronic inflammatory disorders such as sepsis, lung injury, rheumatoid arthritis, and diabetes. Although there are no direct data to demonstrate vagus nerve stimulation's effect in Raynaud's phenomenon, the investigators believe that VNS's success in treating headache and migraine attacks indirectly support its use in Raynaud's phenomenon by its direct effect on vasospasms (narrowing of blood vessels). In fact migraine has been found as a risk factor for the development of Raynaud's phenomenon further supports this notion.

GammaCore is a safe and effective non-drug treatment approved for treating cluster and migraine headaches. It is a patented device that activates the vagus nerve with gentle electrical stimulation. The vagus nerve is an important highway of communication between the brain and many parts of the body, it plays an important role in regulating pain. Noninvasive vagus nerve stimulation with GammaCore is believed to help block the pain signals that cause migraines and cluster headaches. Unlike traditional vagus nerve stimulation therapies, gammaGore stimulates the vagus nerve through the skin at the side of the neck without the need for surgery. This non-invasive method avoids many side effects and inconveniences associated with injectable, inhaled or pill-based medication.

The investigators' goal is to test the possibility that noninvasive vagus nerve stimulation using gammaCore may be an effective and well tolerated therapy for Raynaud's phenomenon. The investigators aim to gain a fundamental understanding of the role of noninvasive vagus nerve stimulation as a potential therapy for Raynaud's phenomenon, a truly unmet medical need.

ELIGIBILITY:
Inclusion Criteria:

• Clinical Diagnosis of Primary Raynaud's Phenomenon

Exclusion Criteria:

* Less than 18 years of age
* Pregnant women
* Current smokers
* Have Digital ulcers
* Diagnosed Pulmonary hypertension
* Currently on vasodilators (i.e. Phosphodiesterase type 5 inhibitors, prostacyclin, nitroglycerine, or other nitric oxide derivatives)
* Currently on Calcium Channel Blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bashar Kahaleh, MD, Principal Investigator — University of Toledo
Locations (1):
- Unversity of Toledo Medical Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garner R, Kumari R, Lanyon P, Doherty M, Zhang W. Prevalence, risk factors and associations of primary Raynaud's phenomenon: systematic review and meta-analysis of observational studies. BMJ Open. 2015 Mar 16;5(3):e006389. doi: 10.1136/bmjopen-2014-006389. PMID 25776043
- [Background] Brand FN, Larson MG, Kannel WB, McGuirk JM. The occurrence of Raynaud's phenomenon in a general population: the Framingham Study. Vasc Med. 1997 Nov;2(4):296-301. doi: 10.1177/1358863X9700200404. PMID 9575602
- [Background] Merkel PA, Herlyn K, Martin RW, Anderson JJ, Mayes MD, Bell P, Korn JH, Simms RW, Csuka ME, Medsger TA Jr, Rothfield NF, Ellman MH, Collier DH, Weinstein A, Furst DE, Jimenez SA, White B, Seibold JR, Wigley FM; Scleroderma Clinical Trials Consortium. Measuring disease activity and functional status in patients with scleroderma and Raynaud's phenomenon. Arthritis Rheum. 2002 Sep;46(9):2410-20. doi: 10.1002/art.10486. PMID 12355489
- [Background] Matucci-Cerinic M, Kahaleh B, Wigley FM. Review: evidence that systemic sclerosis is a vascular disease. Arthritis Rheum. 2013 Aug;65(8):1953-62. doi: 10.1002/art.37988. No abstract available. PMID 23666787
- [Background] Ennis H, Anderson ME, Wilkinson J, Herrick AL. Calcium channel blockers for primary Raynaud's phenomenon. Cochrane Database Syst Rev. 2014 Jan 30;(1):CD002069. doi: 10.1002/14651858.CD002069.pub4. PMID 24482037
- [Background] Coleiro B, Marshall SE, Denton CP, Howell K, Blann A, Welsh KI, Black CM. Treatment of Raynaud's phenomenon with the selective serotonin reuptake inhibitor fluoxetine. Rheumatology (Oxford). 2001 Sep;40(9):1038-43. doi: 10.1093/rheumatology/40.9.1038. PMID 11561116
- [Background] Pauling JD, Shipley JA, Harris ND, McHugh NJ. Use of infrared thermography as an endpoint in therapeutic trials of Raynaud's phenomenon and systemic sclerosis. Clin Exp Rheumatol. 2012 Mar-Apr;30(2 Suppl 71):S103-15. Epub 2012 May 30. PMID 22691218
- [Background] James PB. Cooling patterns in Raynaud's phenomenon and allied peripheral vascular disorders. Br J Surg. 1968 Nov;55(11):860. No abstract available. PMID 5686991
- [Background] Zaproudina N, Varmavuo V, Airaksinen O, Narhi M. Reproducibility of infrared thermography measurements in healthy individuals. Physiol Meas. 2008 Apr;29(4):515-24. doi: 10.1088/0967-3334/29/4/007. Epub 2008 Apr 9. PMID 18401069
- [Background] Pauling JD, Shipley JA, Raper S, Watson ML, Ward SG, Harris ND, McHugh NJ. Comparison of infrared thermography and laser speckle contrast imaging for the dynamic assessment of digital microvascular function. Microvasc Res. 2012 Mar;83(2):162-7. doi: 10.1016/j.mvr.2011.06.012. Epub 2011 Jul 1. PMID 21763703
- [Background] Schlager O, Gschwandtner ME, Herberg K, Frohner T, Schillinger M, Koppensteiner R, Mlekusch W. Correlation of infrared thermography and skin perfusion in Raynaud patients and in healthy controls. Microvasc Res. 2010 Jul;80(1):54-7. doi: 10.1016/j.mvr.2010.01.010. Epub 2010 Feb 6. PMID 20144625
- [Background] Johnson RL, Wilson CG. A review of vagus nerve stimulation as a therapeutic intervention. J Inflamm Res. 2018 May 16;11:203-213. doi: 10.2147/JIR.S163248. eCollection 2018. PMID 29844694
- [Background] Silberstein SD, Calhoun AH, Treppendahl C, Dodick DW, Rapoport AM, Mamidi A, Vargas P, Ebert TH, Tepper SJ. The emerging role of gammaCore(R) in the management of cluster headache: expert panel recommendations. Am J Manag Care. 2017 Nov;23(17 Suppl):S326-S333. PMID 29144718
- See also: Safety information on the gammaCore Sapphire device. — https://gammacore.com/prescribing-gammacore/clinical-safety/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 enrolled
Groups:
- gammaCore: randomized to active treatment
- Sham Device Group: randomized to receive sham device first half of treatment window then switch to gammaCore
Period: Overall Study
Arm/Group | gammaCore | Sham Device Group
Started | 6 | 0 (Unable to locate study records for the Sham Group; unable to confirm how many, if any, were randomized to this arm)
Completed | 6 | 0 (Unable to locate study records for the Sham Group; unable to confirm how many, if any, were randomized to this arm)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Unable to locate study records for the Sham Group; unable to confirm how many, if any, were randomized to this arm
Groups:
- Sham Device Group: randomized to receive sham device first half of treatment window then switch to active treatment
- Total: Total of all reporting groups
Arm/Group | gammaCore | Sham Device Group | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 6 |  | 6
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 |  | 6
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 2 |  | 2
  White | 4 |  | 4
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Temperature in 4 Digits
Description: Temperature measured by infrared thermography
Time Frame: Visit 1 which is Week -4 (Screening) to Visit 2 which is Week 0 (Randomization)
Population: Unable to locate study records for the Sham Group; unable to confirm how many, if any, were randomized to this arm
Measure: Mean (Standard Deviation); unit: degree centigrade
Arm/Group | gammaCore | Sham Device Group
Number analyzed (Participants) | 6 | 0
degree centigrade
  baseline right digit visit 1 | 29.48 (2.43) |
  baseline right digit 2 visit 1 | 28.53 (4.36) |
  baseline right digit 3 visit 1 | 28.70 (4.57) |
  baseline right digit 4 visit 1 | 28.88 (4.49) |
  baseline left digit visit 1 | 29.43 (1.89) |
  baseline left digit 2 visit 1 | 28.53 (4.04) |
  baseline left digit 3 visit 1 | 28.15 (3.87) |
  baseline left digit 4 visit 1 | 28.23 (3.99) |
  right digit, 1 minute, visit 1 | 23.73 (1.51) |
  right digit 2, 1 minute, visit 1 | 20.40 (1.86) |
  right digit 3, 1 minute, visit 1 | 20.30 (1.80) |
  right digit 4,1 minute, visit 1 | 19.85 (1.56) |
  left digit, 1 minute, visit 1 | 23.88 (1.29) |
  left digit 2, 1 minute, visit 1 | 20.13 (1.52) |
  left digit 3, 1 minute, visit 1 | 19.85 (1.41) |
  left digit 4, 1 minute, visit 1 | 19.50 (1.19) |
  right digit, 5 minuets, visit 1 | 24.83 (1.50) |
  right digit 2, 5 minuets, visit 1 | 22.18 (2.92) |
  right digit 3, 5 minutes, visit 1 | 22.40 (3.57) |
  right digit 4, 5 minutes, visit 1 | 22.50 (3.95) |
  left digit, 5 minutes, visit 1 | 25.33 (1.29) |
  left digit 2, 5 minutes, visit 1 | 22.75 (4.22) |
  left digit 3, 5 minutes, visit 1 | 22.75 (4.54) |
  left digit 4, 5 minutes, visit 1 | 23.23 (5.36) |
  right digit , 10 minutes, visit 1 | 25.33 (1.61) |
  right digit 2, 10 minutes, visit 1 | 22.73 (3.12) |
  right digit 3, 10 minutes, visit 1 | 22.90 (3.64) |
  right digit 4, 10 minutes, visit 1 | 22.83 (3.36) |
  left digit , 10 minutes, visit 1 | 26.00 (1.77) |
  left digit 2, 10 minutes, visit 1 | 23.20 (3.95) |
  left digit 3, 10 minutes, visit 1 | 23.03 (4.00) |
  left digit 4, 10 minutes, visit 1 | 23.28 (4.35) |
  right digit, 15 minutes, visit 1 | 25.93 (1.95) |
  right digit 2, 15 minutes, visit 1 | 23.85 (3.58) |
  right digit 3, 15 minutes, visit 1 | 24.80 (4.56) |
  right digit 4, 15 minutes, visit 1 | 24.25 (4.35) |
  left digit, 15 minutes, visit 1 | 26.33 (2.64) |
  left digit 2, 15 minutes, visit 1 | 24.78 (4.79) |
  left digit 3, 15 minutes, visit 1 | 24.30 (4.96) |
  left digit 4, 15 minutes, visit 1 | 24.63 (5.28) |
  right digit, 20 minutes, visit 1 | 26.18 (2.65) |
  right digit 2, 20 minutes, visit 1 | 24.10 (3.96) |
  right digit 3, 20 minutes, visit 1 | 24.65 (4.52) |
  right digit 4, 20 minutes, visit 1 | 24.38 (4.43) |
  left digit, 20 minutes, visit 1 | 26.83 (3.32) |
  left digit 2, 20 minutes, visit 1 | 24.55 (4.64) |
  left digit 3, 20 minutes, visit 1 | 24.38 (4.88) |
  left digit 4 20 minutes, visit 1 | 24.53 (4.97) |
  baseline right digit, visit 2 | 29.78 (2.19) |
  baseline right digit 2, visit 2 | 28.75 (3.13) |
  baseline right digit 3, visit 2 | 28.08 (3.25) |
  baseline right digit 4, visit 2 | 27.85 (3.60) |
  baseline left digit, visit 2 | 29.50 (2.46) |
  baseline left digit 2, visit 2 | 28.08 (3.37) |
  baseline left digit 3, visit 2 | 28.03 (3.58) |
  baseline left digit 4, visit 2 | 27.75 (3.66) |
  1 minute, right digit, visit 2 | 24.15 (1.28) |
  1 minute, right digit 2, visit 2 | 19.95 (1.34) |
  1 minute, right digit 3, visit 2 | 19.85 (1.46) |
  1 minute, right digit 4, visit 2 | 19.35 (1.32) |
  1 minute, left digit, visit 2 | 23.80 (1.57) |
  1 minute, left digit 2, visit 2 | 19.80 (1.28) |
  1 minute, left digit 3, visit 2 | 19.75 (1.24) |
  1 minute, left digit 4, visit 2 | 19.18 (0.82) |
  5 minutes, right digit, visit 2 | 25.60 (1.10) |
  5 minutes, right digit 2, visit 2 | 20.23 (1.23) |
  5 minutes, right digit 3, visit 2 | 20.05 (0.83) |
  5 minutes, right digit 4, visit 2 | 19.75 (0.54) |
  5 minutes, left digit, visit 2 | 24.73 (1.01) |
  5 minutes, left digit 2, visit 2 | 20.43 (0.96) |
  5 minutes, left digit 3, visit 2 | 20.20 (0.82) |
  5 minutes, left digit 4, visit 2 | 20.20 (0.94) |
  10 minutes, right digit, visit 2 | 25.58 (0.78) |
  10 minutes, right digit 2, visit 2 | 20.90 (1.68) |
  10 minutes, right digit 3, visit 2 | 20.53 (0.98) |
  10 minutes, right digit 4, visit 2 | 20.63 (0.98) |
  10 minutes, left digit, visit 2 | 24.85 (0.90) |
  10 minutes, left digit 2, visit 2 | 22.78 (4.23) |
  10 minutes, left digit 3, visit 2 | 22.68 (4.23) |
  10 minutes, left digit 4, visit 2 | 23.25 (5.17) |
  15 minutes, right digit, visit | 25.40 (0.94) |
  15 minutes, right digit 2, visit | 22.50 (4.08) |
  15 minutes, right digit 3, visit | 22.68 (3.89) |
  15 minutes, right digit 4, visit | 22.85 (3.84) |
  15 minutes, left digit, visit 2 | 25.60 (2.60) |
  15 minutes, left digit 2, visit 2 | 23.28 (4.46) |
  15 minutes, left digit 3, visit 2 | 23.35 (4.83) |
  15 minutes, left digit 4, visit 2 | 23.78 (5.16) |
  20 minutes, right digit, visit 2 | 25.45 (1.33) |
  20 minutes, right digit 2, visit 2 | 22.30 (3.05) |
  20 minutes, right digit 3, visit 2 | 22.35 (2.63) |
  20 minutes, right digit 4, visit 2 | 22.55 (2.63) |
  20 minutes, left digit, visit 2 | 25.53 (2.76) |
  20 minutes, left digit 2, visit 2 | 23.00 (3.29) |
  20 minutes, left digit 3, visit 2 | 23.10 (3.64) |
  20 minutes, left digit 4, visit 2 | 23.45 (3.79) |

2. Secondary Outcome: Condition Scores
Description: The Raynaud's Condition Score is on a scale of 0 to 10 with "0" being no difficulty, "10" being extreme difficulty.
Time Frame: n/a - No data was collected.
Population: No data was collected. Diary would have been collected at Week +4 but no subjects reached this time point due to study termination prior to this visit.
Arm/Group | gammaCore | Sham Device Group
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Response Rates
Description: Observe response rates in an open label fashion after subjects randomized to the sham device are transitioned to the gammaCore nVNS device.
Time Frame: n/a - No data was collected. The transition from sham device to open label gammaCore nVNS device would not have occurred until Week +4. No subject reached Week 4 due to study being terminated prior to this visit.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Visit 1 which is Week -4 (Screening) to Visit 2 which is Week 0 (Randomization)
Description: Unable to locate study records for the Sham Group; unable to confirm how many, if any, were randomized to this arm
Groups:
- gammaCore: randomized to active treatment the study was abruptly terminated due to the sponsor's financial problems
Arm/Group | gammaCore | Sham Device Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 0/6 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03869008/Prot_SAP_002.pdf